CLINICAL TRIAL: NCT03361358
Title: Identification of MTAP Deletion in Archival Tumor Tissue: A Pre-Screening Study in Subjects With Advanced Solid Tumors or Lymphoma
Brief Title: Pre-Screening Study to Identify MTAP Loss in Advanced Solid Tumors or Lymphoma
Status: Completed | Type: Observational
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AG270-PS-001
Record Dates: First submitted 2017-11-16; First posted 2017-12-04 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Advanced Solid Tumors; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archived tumor samples will be collected and stored for an unlimited amount of time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify subjects with advanced solid tumors or lymphoma in which the methylthioadenosine phosphorylase (MTAP) protein has been lost.

DETAILED DESCRIPTION:
Study AG270-PS-001 is a pre-screening study to identify subjects with advanced solid tumors or lymphoma in which the MTAP protein has been lost. Subjects whose tumor tissue has lost the MTAP protein may be considered for future enrollment into a Phase 1 clinical study of an experimental drug, AG-270, that is designed to inhibit the growth of tumors lacking this protein.

Identification of the loss of MTAP will rely solely on the evaluation of archival tumor tissue samples by IHC. This study is therefore non-interventional

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years of age.
2. Have a histologically confirmed diagnosis of an advanced solid tumor (other than a primary CNS malignancy) or lymphoma.
3. Have archival tumor tissue that can be provided for assessment of MTAP deletion status.
4. Have given written informed consent to participate in this study.

Exclusion Criteria:

1. Have a primary CNS malignancy (eg, GBM).
2. Have a medical or psychological condition deemed by the Investigator likely to interfere with the subject's ability to give informed consent or participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects appropriate for this study will be identified by the Investigators at the study sites based on their clinical judgment. This study may be conducted in subjects who are not currently eligible for an experimental therapy, recognizing that determination of the tumor's MTAP status could be useful in making future decisions about options for treatment.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Determination of MTAP status in tumors | From initiation of the Pre-Screen study until the Phase 1 study of AG-270 is activated at each study site, up to 9 months
  Number of tumor tissue samples found to have or not have MTAP deletion, as assessed by IHC

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Boston, MA, Boston, Massachusetts
  - Nashville, TN, Nashville, Tennessee
- Barcelona, Spain, Barcelona, Spain